CLINICAL TRIAL: NCT05150392
Title: An Open-labelled Clinical Trial,to Evaluate the Immunity Persistence of the Single-dose Primary Immunization of Live Attenuated Varicella Vaccine on Different Time Points,and the Safety and Immunogenicity After the Booster Immunization
Brief Title: An Open-labelled Clinical Trial of Live Attenuated Varicella Vaccines to Evaluate the Immunity Persistence After Primary Immunization and Safety and Immunogenicity After the Booster Immunization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VZV-3002-1
Record Dates: First submitted 2021-11-22; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Booster immunization 1 year after primary immunization (Experimental): Subjects C0001-C0400 except C0243 received 1 dose of booster immunization 1 year after primary immunization.
  Interventions: Biological: Investigational live attenuated varicella vaccine
- Booster immunization 2 year after primary immunization (Experimental): Subjects C0401-C0800 except C0556 received 1 dose of booster immunization 2 years after primary immunization.
  Interventions: Biological: Investigational live attenuated varicella vaccine
- Booster immunization 3 year after primary immunization (Experimental): Subjects C0801-C1197 received 1 dose of booster immunization 3 years after primary immunization.
  Interventions: Biological: Investigational live attenuated varicella vaccine

INTERVENTIONS:
Biological: Investigational live attenuated varicella vaccine — The investigational vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.And the live varicella-zoster virus in 0·5 mL of sucrose, sodium glutamate,sodium chloride,potassium chloride,sodium dihydrogen phosphate, potassium dihydrogen phosphate and injection water per injection

SUMMARY:
This is an open-labelled clinical trial of live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd .The purpose of this study is to evaluate the immunity persistence of the single-dose primary immunization of live attenuated varicella vaccine on different time points ,and the safety and immunogenicity after the booster immunization

DETAILED DESCRIPTION:
This study is an open-labelled phase Ⅲ clinical trial.The experimental vaccine manufactured by Sinovac(Dalian) Vaccine Technology Co., Ltd.A total of 1195 subjects who received vaccine in the phase Ⅲ lot-consistency clinical trial were be enrolled .All subjects except C0243 and C0556 were divided into 3 groups according to the order of study number.Subjects in 3 groups received a booster immunization of live attenuated varicella vaccines 1 year,2 years and 3 years after primary immunization,respectively.About 3.0ml of venous blood was collected from each enrolled subject at pre-booster immunization,30 days after booster immunization and the serum was separated for neutralizing antibody detection.The antibody levels were used to evaluate the immunity persistence and immunogenicity after booster immunization of live attenuated varicella vaccines .

ELIGIBILITY:
Inclusion Criteria:

* Received one dose live attenuated varicella vaccine in the phase Ⅲ lot-consistency clinical trial;
* Guardian(s) of the volunteer should be capable of understanding the written - consent form, and such form should be signed before the children being included into this study.

Exclusion Criteria:

* Received one dose live attenuated varicella vaccine at the end of the phase Ⅲ lot-consistency clinical trial;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1193 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-seroconversion rate of antibody | 1 year after primary immunization
  seroconversion rates of antibody 1 year after primary immunization
Immunogenicity index-seroconversion rate of antibody | 2 years after primary immunization
  seroconversion rates of antibody 2 years after primary immunization
Immunogenicity index-seroconversion rate of antibody | 3 years after primary immunization
  seroconversion rates of antibody 3 years after primary immunization
Immunogenicity index-Seroconversion rate of antibody | 30 days after booster immunization
  Seroconversion rate of the neutralizing antibody 30 days after booster immunization
Immunogenicity index-seropositivity rate of antibody | 30 days after booster immunization
  Seropositivity rate of antibody 30 days after booster immunization

SECONDARY OUTCOMES:
Immunogenicity index-Seropositivity rate of antibody | Before the booster dose immunization
  Seropositivity rate of antibody before booster immunization
Immunogenicity index-GMT of the antibody | Before the booster dose immunization
  GMT of the antibody before booster immunization
Immunogenicity index- GMT of the antibody | 30 days after booster immunization
  GMT of the antibody 30 days after booster immunization
Immunogenicity index- GMI of the antibody | 30 days after booster immunization
  GMI of the antibody 30 days after booster immunization
Safety index-Incidence of solicited local or systemic AE | within 14 days after vaccination
  Incidence of solicited local or systemic AE within 14 days after vaccination
Safety index-Incidence of local or systemic AE | within 30 days after vaccination
  Incidence of local or systemic AE within 30 days after vaccination
Safety index-Incidence of SAE | within 30 days after vaccination
  Incidence of SAE within 30 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Xia, Master, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Xiangfu County Center for Disease Control and Prevention, Kaifeng, Henan, China